CLINICAL TRIAL: NCT03920124
Title: Exploring the Feasibility and Effectiveness of Minimal-equipment High-intensity Interval Exercise (HIIE) Interventions in Bronchiectasis Patients
Brief Title: Feasibility of Interval Exercise in Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: United Lincolnshire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 180901
Record Dates: First submitted 2018-10-05; First posted 2019-04-18 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: This will be a pragmatic feasibility study of a single case group. However, examination of acute responses to different step and walk-based interval exercise types will follow a randomised, counter-balanced (repeated-measures) design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High intensity interval exercise (Experimental): Completion of four separate step and walk-based high intensity interval exercise sessions, followed by completion of six week unsupervised (at home) high intensity interval exercise intervention
  Interventions: Other: Step and walk-based high intensity interval exercise

INTERVENTIONS:
Other: Step and walk-based high intensity interval exercise — Four hospital-based trials will include two step-based (3 x 20 sec with 120 sec rest, or 3 x 60 sec with 60 sec rest) and two walking-based (e.g. 3 x 60 sec with 60 sec rest or 3 x 180 sec with 180 sec rest) interval exercise protocols, in a randomised and counterbalanced order.
  Unsupervised (At home) exercise intervention will incorporate patients' preferred stair and/or walking-based interval exercise (from those completed during hospital trials). Initially patients will complete their chosen protocol three days per week, and then gradually progress exercise load (i.e. reps, work-to-rest ratio, and/or sessions per week) as appropriate, to a maximum of 6 x 60 sec stepping / 5 x 180 sec walking, five times per week (i.e. maximum of ~30 min daily or ~150 min weekly).

SUMMARY:
Research to date suggests that encouraging increased physical activity and exercise engagement may be an effective way to improve symptoms, fitness, quality of life, and reduce time spent in hospital for bronchiectasis sufferers. However, relatively few patients continue to engage with exercise programs that are of benefit to their health and symptoms. Barriers to exercise are thought to include time constraints and the use of specialist equipment (e.g. cycle ergometers) which may not be available or accessible in the home (or hospital) setting. With these points in mind, there is growing interest in brief, relatively intense, interval exercise interventions for chronic lung disease sufferers as they require minimal equipment and may more easily translate back into the home setting. Of the types of approach this might include, both stair-based and walk-based interval exercise appear to be relatively safe, practical, and time-efficient ways to improve physical fitness and quality of life in previously untrained and clinical populations. However, the feasibility and effectiveness of their use by chronic lung disease patients, particularly those with bronchiectasis, is yet to be properly examined. The investigators therefore intend to recruit 10 bronchiectasis patients to explore the feasibility and effectiveness of minimal-equipment interval exercise interventions in this population. More specifically, the investigators would like to observe patients' acute physical and perceptual responses to four different step and walk-based protocols which have been established for other clinical populations. The investigators also wish to explore whether these protocols are engaged with, and enjoyed, during a six week unsupervised exercise intervention (in the home), as well as the effects of this six week unsupervised exercise period on physical fitness. This project will hopefully make a valuable contribution to the limited research to have examined the real-world application and impact of interval-type exercise interventions on exercise behaviour, health, and symptoms in bronchiectasis sufferers.

DETAILED DESCRIPTION:
Baseline testing (Visit 1) Having completed informed consent and screening, participants will be invited to complete a hospital-based baseline physiological testing session. The usual care of this participant group means that a clinical assessment of condition severity and associated spirometry measures (e.g. peak flow, forced vital capacity) will have already been completed which will be included in the study data. If this is not the case, then a member of the patient's usual care team (which may include members of the research team) will collect these baseline measures. Baseline physiological assessment will then be completed, including a self-paced six minute walk test (6MWT); an Isometric Quadriceps Strength Test (IQST); and an incremental, externally paced, symptom-limited Chester Step Test (CST ). Peak values for cardiorespiratory measures (i.e. heart rate, oxygen consumption and saturation, minute ventilation) will be established by way of clinically validated metabolic cart, oximeter and facemask applied during the incremental CST. Each of these tests will be delivered in the stated order across a 60 minute period, with each test followed by at least 5 minutes of rest to allow for adequate recovery and instruction.

Acute high-intensity interval exercise trials (Visits 2-5) Four subsequent hospital-based (supervised) trials will require participants to complete differing formats of step-based or walking-based HIIE, in a randomised order established by an online random sequence generator. Mean and peak values for cardiorespiratory responses (i.e. heart rate, oxygen consumption, minute ventilation) will be established by way of clinically validated metabolic cart and face-mask applied for the duration of each protocol. Whilst the same format of each HIIE session will prescribed to each participant, their completion of each work and rest period (and the duration of these) will be subject to symptom limitation (i.e. they will be permitted to shorten work and/or extend rest periods if symptoms dictate).

Post-HIIE questions will be verbally asked of participants at the end of each exercise session, including;

Did they enjoy this type of exercise? Would they like to try this exercise at home? Did they feel safe when completing this exercise? What will be the major barrier for them to not try this exercise at home?

In addition to their initial responses, participants will be invited to offer a brief explanation as appropriate. All responses will be recorded by dictaphone and subsequently transcribed by a member of the research team for later analysis.

Unsupervised 6 week high-intensity interval exercise intervention Having completed all acute high-intensity interval exercise trials, participants will then complete 6 weeks of home-based unsupervised exercise, initially incorporating their preferred format of stair and/or walking-based HIIE, three days per week. They will be encouraged to gradually progress exercise load (i.e. repetitions, work-to-rest ratio, and/or sessions per week) to a maximum of 6 x 60 seconds, five times per week (i.e. ~12 minutes total). Measures of physiological status, symptoms and well-being will be logged throughout (i.e. heart rate, dyspnea, respiratory quality of life, anxiety and depression).

Follow-up testing (Visit 6) Upon completion of home-based unsupervised exercise intervention, baseline physiological assessments will be repeated in the hospital setting. This will again include a self-paced MWT; an IQS test; and an incremental, externally paced, symptom-limited CST. Peak values for cardiorespiratory measures (i.e. heart rate, oxygen consumption, minute ventilation) will be established by way of clinically validated metabolic cart and facemask applied during the incremental CST. Each of these tests will be delivered in the stated order across a 60 minute period, with each test followed by at least 15 minutes of rest to allow for adequate recovery and instruction.

Following a similar approach to pre-intervention testing, post-intervention questions will be verbally asked of participants at the end of the follow up testing session, including; Did they enjoy this exercise intervention? Would they like to continue these types of exercise at home? Did they feel safe when completing these exercises at home? What will be the major barrier for them to not continue these types of exercise at home? What changes would make continuing this type of exercise more appealing to them?

In addition to their initial responses, participants will be invited to offer a brief explanation as appropriate. All responses will be recorded by dictaphone and subsequently transcribed by a member of the research team for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (i.e. >18 years)
* Clinical diagnosis of non-cystic fibrosis bronchiectasis.
* Registered/treated as an inpatient or outpatient with the United Lincolnshire NHS Trust
* Capable of giving informed consent.
* Deemed eligible for pulmonary rehabilitation (including exercise) by clinical specialist, specialist nurse, or respiratory physiotherapist.
* Has not met national guidelines for exercise engagement during the preceding 3 months (i.e. completing at least 150 minutes of moderate aerobic activity or 75 minutes of vigorous aerobic activity each week).

Exclusion Criteria:

* Inability or unwillingness to sign informed consent;
* Outside of stated age range (i.e. <18 years);
* Pregnant;
* Suffering from any major co-morbidity known to impair exercise tolerance (i.e. heart failure/disease, diabetes, neuromuscular and/or musculoskeletal disease or injury) or another factor considered as a contraindication to clinical exercise testing by clinical specialist respiratory physiotherapist;
* Has met national guidelines for exercise engagement during the previous 3 months (i.e. completing at least 150 minutes of moderate aerobic activity or 75 minutes of vigorous aerobic activity each week)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Completion rate | Week 11 (i.e. visit 6)
  Completion rate (%) for each type of interval exercise protocol administered
Emergent adverse events | Week 11 (i.e. visit 6)
  Number of adverse events (count) during high-intensity interval exercise protocols

SECONDARY OUTCOMES:
Heart rate | Captured at Baseline and throughout each interval exercise bout during visits 2, 3, 4, 5 and 6 (i.e. weeks 1, 2, 3, 4, 5 and 11)
  Mean and peak heart rate values (beats per minute)
Oxygen consumption | Captured at Baseline and throughout each interval exercise bout during visits 2, 3, 4, 5 and 6 (i.e. weeks 1, 2, 3, 4, 5 and 11)
  Mean and peak oxygen consumption values (millilitres per kilogram per minute)
Minute ventilation | Captured at Baseline and throughout each interval exercise bout during visits 2, 3, 4, 5 and 6 (i.e. weeks 1, 2, 3, 4, 5 and 11)
  Mean and peak minute ventilation values (litres per minute)
Respiratory frequency | Captured at Baseline and throughout each interval exercise bout during visits 2, 3, 4, 5 and 6 (i.e. weeks 1, 2, 3, 4, 5 and 11)
  Mean and peak respiratory frequency values (breaths per minute)
Oxygen saturation | Captured at Baseline and throughout each interval exercise bout during visits 2, 3, 4, 5 and 6 (i.e. weeks 1, 2, 3, 4, 5 and 11)
  Mean and peak oxygen saturation values (% SpO2)
Perceived fatigue during interval exercise | Captured during the final 3 min of interval exercise bouts and the first 3 mins of the post-exercise recovery phase
  Fatigue [Borg CR 0-10 Scale]
Perceived breathlessness during interval exercise | Captured during the final 3 min of interval exercise bouts and the first 3 mins of the post-exercise recovery phase
  Perceived Breathlessness [Borg CR 0-10 Scale]
Affect/Pleasure response to interval exercise | Captured during the final 3 min of interval exercise bouts and the first 3 mins of the post-exercise recovery phase
  Affect/Pleasure [Feeling Scale -5 to +5 Score]
Six-Minute Walk Test Performance | Change from Baseline to visit 6 (i.e. weeks 1 to 11)
  Six-Minute Walk Test (distance in meters)
Chester Step Test Performance | Change from Baseline to visit 6 (i.e. weeks 1 to 11)
  Chester Step Test (final step rate in steps per minute)
Quadriceps Strength | Change from Baseline to visit 6 (i.e. weeks 1 to 11)
  Isometric Quadriceps Strength Test (peak force [kg/N])
Patient perceptions of interval exercise protocols | Captured during visits 2, 3, 4, 5 and 6 (i.e. weeks 2, 3, 4, 5 and 11)
  Interview questions
EuroQoL (EQ-5D-5L) questionnaire for health-related quality of life | Captured at Baseline and then weekly during intervention period (i.e. weeks 1, 6, 7, 8, 9, 10 and 11)
  EuroQoL (EQ-5D-5L) questionnaire for health-related quality of life: 5 Dimensions - Mobility, self-care, usual activities, pain/discomfort, anxiety/depression including 1 item each with 5 levels
Exacerbations and/or adverse events during interval exercise | Captured at Baseline and then weekly during intervention period (i.e. weeks 1, 6, 7, 8, 9, 10 and 11)
  Event based, patient reported

CONTACTS AND LOCATIONS:
Overall Officials: Danny Taylor, PhD, Principal Investigator — University of Lincoln
Locations (1):
- Lincoln County Hospital Physiotherapy Unity, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No